CLINICAL TRIAL: NCT05199688
Title: A Phase III, Multicenter, Open-Label, Uncontrolled Study To Evaluate Pharmacokinetics, Efficacy, Safety, Tolerability, And Pharmacodynamics Of Satralizumab In Pediatric Patients With AQP4 Antibody Positive Neuromyelitis Optica Spectrum Disorder (NMOSD)
Brief Title: A Study To Evaluate Pharmacokinetics, Efficacy, Safety, Tolerability, And Pharmacodynamics Of Satralizumab In Pediatric Patients With Aquaporin-4 Antibody Positive Neuromyelitis Optica Spectrum Disorder (NMOSD)
Acronym: SAkuraSun
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WN41733; 2019-004092-39 (EudraCT Number); 2023-507817-85-00 (EU CTIS Number)
Record Dates: First submitted 2021-12-03; First posted 2022-01-20 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Neuromyelitis Optica Spectrum Disorder; NMOSD
MeSH Terms: conditions — Neuromyelitis Optica | interventions — satralizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort 1: Participants with body weight ≥10kg to <20kg (Experimental): Satralizumab will be administered SC Q6W in a cohort of at least 2 evaluable patients
  Interventions: Drug: Satralizumab
- Cohort 2 Participants with body weight ≥20kg to <40kg (Experimental): Satralizumab will be administered SC at Weeks 0, 2, 4, and Q4W thereafter.
  Interventions: Drug: Satralizumab
- Cohort 3 Participants with body weight ≥40kg (Experimental): Satralizumab will be administered SC at Weeks 0, 2, 4, and Q4W thereafter.
  Interventions: Drug: Satralizumab

INTERVENTIONS:
Drug: Satralizumab — Participants will receive satralizumab treatment for a minimum of 48 weeks and then will have the opportunity to enter an optional satralizumab extension (OSE) period.

SUMMARY:
This study will primarily evaluate the pharmacokinetics of satralizumab in pediatric patients aged 2-11 years with anti-aquaporin-4 (AQP4) antibody seropositive neuromyelitis optica spectrum disorder (NMOSD). Efficacy, safety, tolerability, and pharmacodynamics will be evaluated in a descriptive manner, given the small number of patients who will be enrolled in this study.

ELIGIBILITY:
Inclusion Criteria:

* Age at screening 2-11 years, inclusive
* Body weight at screening >=10 kg
* For female patients of childbearing potential (postmenarchal): agreement to either remain completely abstinent (refrain from heterosexual intercourse) or to use a reliable means of contraception
* Diagnosed as having NMOSD with AQP4 antibody seropositive status as defined by the Wingerchuk 2015 criteria Clinical evidence of at least one documented attack (including first attack) in the last year prior to screening
* Neurological stability for >=30 days prior to both screening and baseline
* Expanded Disability Status Scale (EDSS) 0 to 6.5
* For patients receiving a baseline immunosuppressant treatment and planning to continue on these therapies, treatment must be at stable dose for 4 weeks prior to baseline

Exclusion Criteria:

* Pregnancy or lactation
* Evidence of other demyelinating disease mimicking NMOSD
* Active or presence of recurrent bacterial, viral, fungal, mycobacterial infection, or other infection at baseline
* Evidence of chronic active hepatitis B or C
* Evidence of untreated latent or active tuberculosis (TB)
* Receipt of a live or live-attenuated vaccine within 6 weeks prior to baseline
* History of severe allergic reaction to a biologic agent

Ages: 2 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 8 (Estimated)
Dates: Start 2025-12-31 (Estimated); Primary Completion 2027-03-31 (Estimated); Study Completion 2029-09-12 (Estimated)

PRIMARY OUTCOMES:
Summary of observed serum concentration [Cthrough] of satralizumab | Week 48
Apparent clearance [CL/F] of satralizumab | Week 48
Apparent volume of distribution [V/F] of satralizumab | Week 48
Area under the concentration-time curve [AUC] of satralizumab | Week 48

SECONDARY OUTCOMES:
Proportion of relapse-free patients by Week 48 | Week 48
Annualized relapse rate (ARR), defined as the average number of relapses for each year of the study | Week 48
Time to first relapse (TFR) after randomization, defined as the time from randomization until the first occurrence of relapse, as determined by the investigator | Week 48
Time to relapse requiring rescue therapy | Week 48
Change from baseline in Expanded Disability Status Scale (EDSS) at Weeks 24 and 48 | Baseline, Week 24, Week 48
Change from baseline in visual acuity at Weeks 24 and 48 | Baseline, Week 24, Week 48
Change from baseline in FACES Pain Rating Scale at Weeks 24 and 48 | Baseline, Week 24, Week 48
Change from baseline in EuroQol 5-Dimension, Youth (EQ-5D-Y) score and its proxy at Weeks 24 and 48 | Baseline, Week 24, Week 48
Incidence and severity of adverse events | Week 48

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (10):
- Children's Hospital Colorado., Denver, Colorado, United States
- Argentina (2):
  - Hospital de Pediatría S.A.M.I.C.- Prof. Dr. Juan P. Garrahan, Ciudad Autonoma Buenos Aires
  - Clinica Universitaria Reina Fabiola, Córdoba
- Centre Hospitalier Universitaire de Bicêtre, Le Kremlin-Bicêtre, France
- Italy (2):
  - IRCCS Ospedale Pediatrico Bambino Gesù - INCIPIT - PIN, Rome, Lazio
  - Fondazione Istituto Neurologico Mondino IRCCS, Pavia, Lombardy
- Grupo Medico Camino, DF, Mexico CITY (federal District), Mexico
- Uniwersyteckie Centrum Kliniczne, Gda?sk, Poland
- Kocaeli University Research and Application Hospit, Kocaeli, Turkey (Türkiye)
- Great Ormond Street Hospital for Children, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
For eligible studies, qualified researchers may request access to individual patient level clinical data. See Roche's commitment to transparency of clinical study information here: https://go.roche.com/data_sharing